CLINICAL TRIAL: NCT00222976
Title: Oral vs Rectal Administration of Naproxen for Post-Vaginal Perineal Pain Control: A Randomized Clinical Trial
Brief Title: Oral vs Rectal Admin of Naproxen for Post-Vag Perineal Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bio-REB 05-96
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Post-Vaginal Delivery Perineal Pain
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): A Naproxen PO + placebo PR
  Interventions: Drug: Naproxen
- 2 (Experimental): B Placebo PO + Naproxen PR
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — Treatment allocation either A Naproxen PO + placebo PR or B Placebo PO + Naproxen PR

SUMMARY:
The primary objective of this study is to determine whether the route of administration of naproxen (either by mouth or rectally) influences post-vaginal delivery perineal pain control.

DETAILED DESCRIPTION:
Postpartum perineal pain is common after vaginal delivery. Naproxen suppositories have been shown to be effective at reducing postpartum perineal pain. To date, no studies have investigated the efficacy of oral naproxen for perineal pain control. Currently, rectal naproxen is used postpartum because of an assumption that there is a "local effect" compared to oral administration. However, this effect has never been documented in the literature.

Principles of pharmacology dictate that the least invasive route of drug administration should be used when two or more routes are equally effective. If oral and rectal naproxen are equally efficacious at controlling post-vaginal delivery perineal pain, then current practice would be challenged.

The primary objective of this study is to determine whether the route of administration of naproxen influences post-vaginal delivery perineal pain control. Pain scores will be measured using a visual analog scale. The secondary outcome measures are three-fold: patient preference of route of administration, medication adverse effects, and additional requests for analgesia. The working hypothesis is that there is no difference in pain control between oral and rectal administration and that patients will prefer the oral route.

ELIGIBILITY:
Inclusion Criteria:

* Potential volunteers who meet all of the following criteria are eligible for this study:

  1. Active labor, whether spontaneous or induced
  2. Age between 18 and 40 years old
  3. Nulliparous
  4. BMI < 40
  5. Single live intrauterine fetus in cephalic presentation
  6. Term gestation (370 weeks to 416 weeks inclusive) as defined by ultrasound or last menstrual period dating
  7. Intrapartum epidural labour analgesia
  8. Written informed consent

Exclusion Criteria:

* Potential volunteers meeting one of more of the following criteria may not be enrolled:

  1. Medical conditions including:

     1. Naproxen, aspirin or other non-steroidal anti-inflammatory drug hypersensitivity
     2. Asthma
     3. Peptic ulcer disease or other inflammatory gastrointestinal disease
     4. Renal, hepatic or cardiac disease
     5. Coagulopathy
     6. Rectal or anal pathology including recent (within 1 month) rectal bleeding
     7. Prescribed medications including lithium, furosemide, antihypertensives, anticoagulants, aminoglycosides, hydantoins, or sulfonamides
  2. Obstetrical conditions including:

     1. Multiple pregnancy
     2. Extensive perineal trauma (third or fourth degree laceration)
     3. Forceps delivery
     4. Cesarean section delivery
     5. Paracervical or pudendal nerve blocks
     6. Vulval or vaginal hematomas
  3. Nulliparous women not requiring intrapartum epidural labour analgesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
post-vaginal delivery perineal pain scores will be measured using a visual analog scale. | 1 day

SECONDARY OUTCOMES:
patient preference of route of administration | 1 day
medication adverse effects | until completion of study
additional requests for analgesia. | until completion of study

CONTACTS AND LOCATIONS:
Overall Officials: David C Campbell, MD,MSC,FRCPC, Principal Investigator — University of Saskatchewan
Locations (1):
- Department of Anesthesia, Royal University Hospital, University of Saskatchewan, Saskatoon, Saskatchewan, Canada